CLINICAL TRIAL: NCT05230277
Title: OSTEOPATHY IN THE TREATMENT OF IBS SYMPTOMS IN ADULTS: STUDY PROTOCOL FOR A RANDOMIZED CONTROLLED TRIAL
Brief Title: OSTEOPATHY IN THE TREATMENT OF IBS SYMPTOMS IN ADULTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier de Troyes (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TREAT OF IBS SYMPTOMS IN ADULT
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: OSTEOPATHY IN THE TREATMENT OF IBS SYMPTOMS IN ADULTS

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group is defined by the sham osteopathic treatment (SOT) (Placebo Comparator): Patients will receive 3 SOT of 30 minutes each for 2 weeks in a private practice by an experienced osteopath who will receive prior training to optimize the quality of the SOT. The positions of the patient and the practitioner will be the same as in the AOT group
  Interventions: Other: the sham osteopathic treatment
- The experimental group is defined by the active osteopathic treatment (AOT) (Experimental): Patients will receive 3 AOT of 30 minutes each for 2 weeks in a private practice by an experienced osteopath who will receive prior training to optimize the quality of the AOT.
  Interventions: Other: the active osteopathic treatment (AOT)

INTERVENTIONS:
Other: the active osteopathic treatment (AOT) — The AOT will first consist of the application of a visceral technique. The patient will lie on their stomach and the osteopath will touch the patient's abdomen with a wide two-handed grip. The action will consist of following the abdominal tissues in directions where tissue mobility is allowed and occurs without restriction, from the surface to the depth of the abdomen. A change in the elasticity of the colon will then be perceived when the mobility restrictions of the tissues are dissipated. The osteopath will then use a technique on the sacrum according toik-g the procedure described by Attali et al. [8] which consists in mobilizing the sacrum between the iliac bones.
  Arms: The experimental group is defined by the active osteopathic treatment (AOT)
Other: the sham osteopathic treatment — For SOT, the patient will lie on their stomach and the osteopath will use a wide two-handed grip on the patient's abdomen to deliberately mobilize it in an imprecise manner. Next, a technique with no apparent therapeutic effects, the light touch, first described by Licciardone et al. [13] and proposed by others to perform simulated bone manipulations [14], will be applied to the sacrum
  Arms: The experimental group is defined by the sham osteopathic treatment (SOT)

SUMMARY:
Osteopathy is chosen by patients as a treatment for IBS but the evidence for its effectiveness is poor. The purpose of this study is to evaluate the effectiveness of osteopathy for IBS at 1 month follow-up in IBS adults.

DETAILED DESCRIPTION:
a multicenter, two-group parallel, randomized, double-blind, placebo-controlled trial. Inclusion criteria: adult IBS patients (Rome IV criteria) with similar baseline symptom severity, and comparable expectations of active and sham osteopathic treatment before. Treatment group: active osteopathic treatment. Control group: sham osteopathic treatment. Randomization: allocation ratio 1:1. Assessment times: inclusion and baseline assessment (Day-1; Initial visit V0), Day 8, Day 15 and follow-up (1 month and 3 months), treatments (Day 0, Day 8, Day 15). Primary endpoint: Effectiveness at 1 month (response to treatment defined as at least a 50-point reduction in IBS severity on the IBS-symptom severity score). Secondary endpoint: Effectiveness at 3 months (response to treatment) and changes in total IBS quality of life scores up to 3 months. Sample size: 404 individuals to achieve 90% power to detect a 15% difference in treatment response at 1 month between the two groups (20% of patients lost to follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 ans
* IBS patients (defined according to the Rome IV Criteria)
* Moderate symptom severity score on the IBS Symptom Severity Scale (IBS-SSS) (values ranging from 175 to 300).
* Negative colonoscopy within the last 5 years.
* Psychologically fit to provide signed informed consent.
* Agreed to undergo the procedures associated with the study
* Medical insurance

Exclusion Criteria:

* Have not received any osteopathic treatment in the last 12 months
* Chronic inflammatory bowel disease or digestive cancer (even if the disease is in remission)
* Pregnancy
* Planned or expected elective surgery during the study
* Dietary and lifestyle changes in the previous month.
* Use of prohibited concomitant medications in the previous month.
* Inability to understand or cooperate during the study.
* No current participation in a biomedical research trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
The effectiveness (response to treatment) at 1-month follow-up: | 1 month
  It is measured by the IBS symptoms severity score (IBS-SSS) after osteopathic treatment. The IBS-SSS is a validated measure to assess the severity of IBS symptoms, and allows monitoring of the response to treatment.

SECONDARY OUTCOMES:
Effectiveness at 3 months (response to treatment based on the IBS-SSS) and changes in total IBS-Quality Of Life (IBS-QOL) scores up to 3 months. | 3 months
  It is measured by the IBS symptoms severity score (IBS-SSS) after osteopathic treatment. The IBS-SSS is a validated measure to assess the severity of IBS symptoms, and allows monitoring of the response to treatment.
  Changes in total IBS-Quality Of Life (IBS-QOL) scores up to 3 monthsThe IBS-QOL is a self-report measure of quality of life specific to irritable bowel syndrome (IBS) often used to assess the impact of IBS and its treatment.